CLINICAL TRIAL: NCT05100524
Title: The Effect of Motivational Interview for Daily Living Activities on Physical Adjustment and Quality of Life in Elderly People Who Have Had Total Knee Replacement
Brief Title: Motivational Interview for Daily Living Activities in Elderly People Undergoing Total Knee Replacement
Acronym: Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gizem KUBAT BAKIR, Lecturer, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0050
Record Dates: First submitted 2021-09-13; First posted 2021-10-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Motivation; Behavior, Health; Nursing Caries; Nurse's Role
Keywords: motıvatıonal ıntervıew; total knee prosthesıs; old age; quality of life; physical compatibility
MeSH Terms: conditions — Health Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview (Experimental): 8 motivational interviews were conducted with the intervention group.
  Interventions: Other: Motivational interview
- Control Group (Active Comparator): No application was made to increase physical compliance and improve quality of life.
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Motivational interview — The motivational interviewing technique is a client-focused, directive form of counseling to create behavior change. Its main goal is to discover and solve ambivalence. This method is especially useful for people who are reluctant or ambivalent to change.
  Arms: Motivational interview
Other: Ongoing treatment — Patients with total knee replacement receive standard nurse care. Treatment is applied. He does his own exercises at home.
  Arms: Control Group

SUMMARY:
Purpose: In this study, it was aimed to examine the effect of motivational interview on daily living activities on physical adaptation and quality of life in elderly people who underwent total knee replacement.it was aimed to examine the effect of motivational interview on daily living activities on physical adaptation and quality of life in elderly people who underwent total knee replacement.

Design: The research was planned as a pretest, posttest, randomized controlled study in order to determine the effect of the motivational interviews on the life quality and physical activity of old patients.

H1: After total knee replacement, the target for daily living activities is higher than the patients who applied the hand and those who did not.

H2: Patients with targeted daily living activities with total knee replacement begin to get used to it and begin earlier than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 65 and over,
* Having total knee replacement,
* The non-spiritual system (the peasant of the sick),
* A person who can read and write can cope at a level that prevents conversation,
* First time system add-on,
* They are viewed as agreeing to participate in the research.

Exclusion Criteria:

* Neurological (such as dementia) and psychiatric (such as schizophrenia) medical diagnoses that affect cognitive status
* Patients who did not participate in the motivational interviews and who wanted to leave the study were determined.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
The SF-36 Quality of Life Scale | For 3 months
  The SF-36 Quality of Life Scale consists of 8 subgroups and 36 questions. The fourth and fifth questions of the SF-36 scale are yes/no, the other questions are likert type (3, 5 and 6). Items 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, 11d in the scale are calculated by reversing them. The physical and mental summary value of the scale is obtained by adding the weighted scores of the questions containing the sub-scales of the SF-36 quality of life scale. There is no total score. The scores obtained range from zero to one hundred. Zero indicates poor health and 100 indicates good health.
Functional Evaluation Form | For3 months
  The Functional Evaluation Form consists of 8 sections, including maximum walking distance, use of walking aids, getting up from a chair, climbing stairs, working status, daily tasks, transportation and lower extremity care, and each section is self-contained (first four sections are out of 15 points, the remaining four sections are out of 10 points). The highest total score is 100. An increase in the score indicates functional improvement.

CONTACTS AND LOCATIONS:
Overall Officials: GİZEM KUBAT BAKIR, Principal Investigator — GİZEM KUBAT BAKIR
Locations (1):
- Gizem Kubat Bakir, Ataşehir, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Motivational interviewing to increase physical activity in long-term cancer survivors: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/17179870/
- See also: Effectiveness of a motivational interviewing intervention on weight loss, physical activity and cardiovascular disease risk factors: a randomised controlled trial with a 12-month post-intervention follow-up — https://ijbnpa.biomedcentral.com/articles/10.1186/1479-5868-10-40